CLINICAL TRIAL: NCT02376920
Title: CLEAR Registry Study: An Open, 5-year Registry Study to Track Clinical Application of DecisionDx-UM Multigene Assay Results and Associated Patient Outcomes.
Brief Title: 5 Year Registry Study to Track Clinical Application of DecisionDx-UM Assay Results and Associated Patient Outcomes
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: Castle Biosciences Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 2-01
Record Dates: First submitted 2015-02-13; First posted 2015-03-03 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Uveal Melanoma
Keywords: occular melanoma; melanoma of eye; DecisionDx-UM
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Uveal Melanoma is a rare cancer with approximately 3,000 cases diagnosed in the US every year. Nearly half of these experience spread of their cancer outside the eye. The DecisionDx-UM gene expression test classifies an individual's tumor as low risk (class 1) or high risk (class 2) of spreading. This study is being done to collect information about how physicians are using the DecisionDx-UM results to design individual treatment plans. It will also track outcomes or the uveal melanoma population that received DecisionDx-UM testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Uveal Melanoma
* Patients whose physician deems them appropriate for DecisionDx-UM testing
* Patients reasonably able to follow up with enrolling physician at regular intervals for assessment of outcome data

Exclusion Criteria:

* Patients with any other form of cancer

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with uveal melanoma and determined by their treating physician to be appropriate for DecisionDx-UM testing.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2010-03; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
documentation of clinical application of results obtained from DecisionDx-UM multi-gene assay | Approximately 3-6 weeks after biopsy of uveal tumor
  Physician treatment plan with regards to surveillance regimen as well as treatment referral pattern
Time to metastasis | Patients followed for up to 10 years, measurement for metastatic event performed at 6 month intervals

SECONDARY OUTCOMES:
changes in health care costs | Patients followed for up to 10 years at 6 month intervals
  review of health care testing (imaging, laboratory testing) to determine changes in health care costs resulting from DecisionDx-UM testing

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cook, PhD, Principal Investigator — Castle Biosciences Inc.

REFERENCES:
- [Derived] Plasseraud KM, Cook RW, Tsai T, Shildkrot Y, Middlebrook B, Maetzold D, Wilkinson J, Stone J, Johnson C, Oelschlager K, Aaberg TM. Clinical Performance and Management Outcomes with the DecisionDx-UM Gene Expression Profile Test in a Prospective Multicenter Study. J Oncol. 2016;2016:5325762. doi: 10.1155/2016/5325762. Epub 2016 Jun 30. PMID 27446211